CLINICAL TRIAL: NCT05186220
Title: Endocardial Ablation of Ganglionated Plexi Versus Pacemaker Implantation in Patients With Symptomatic Sinus Node Dysfunction
Brief Title: Cardioneuroablation Versus Pacemaker Implantation for the Treatment of Symptomatic Sinus Node Dysfunction
Acronym: DINERVAPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Spanish Society of Cardiology (Other); Hospital Universitario Lucus Augusti (Other)
Responsible Party: Principal Investigator, Carlos Minguito Carazo, Principal Investigator, Cardiology consultant, Electrophysiology fellow, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/307
Record Dates: First submitted 2021-12-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Sinus Node Dysfunction; Sick Sinus Syndrome
Keywords: cardioneuroablation
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioneuroablation (Experimental): After 3D mapping of the surface of the left and right atrium and the superior vena cava (Ensite Navx or Carto system), localization of ganglion plexus (GP) will be performed either anatomically and/or by means of high frequency stimulation (HFS). The anterior and superior right sided GP will always be ablated per protocol. Other GP will be ablated according to interventional electrophysiologist judgement. The endpoint of the ablation procedure will be 1) absence of a vagal response after HFS from the right jugular vein and 2) an increase in at least 10 bpm as compared to baseline.
  Interventions: Procedure: Cardioneuroablation
- Permanent pacemaker implantation (Active Comparator): A dual chamber pacemaker implantation will be performed. The device will be programmed in a AAI-DDDR mode to avoid unnecessary ventricular pacing.
  Interventions: Device: Permanent dual chamber pacemaker implantation

INTERVENTIONS:
Procedure: Cardioneuroablation — After 3D mapping of the surface of the left and right atrium and the superior vena cava (Ensite Navx, Carto), localization of ganglion plexus (GP) will be performed either anatomically and/or by means of high frequency stimulation (HFS). The anterior and superior right sided GP will always be ablated per protocol. Other GP will be ablated according to interventional electrophysiologist judgement. The endpoint of the ablation procedure will be 1) absence of a vagal response after HFS from the right jugular vein and 2) an increase in at least 10 bpm as compared to baseline.
  Other Names: Endocardial ganglion plexus ablation
  Arms: Cardioneuroablation
Device: Permanent dual chamber pacemaker implantation — Under local anesthesia and using a subclavian or cephalic vein approach a dual chamber pacemaker implantation with a lead in the right atrium and a lead in the right ventricle will be performed. The device will be programmed in a AAI-DDDR mode to avoid unnecessary ventricular pacing.
  Arms: Permanent pacemaker implantation

SUMMARY:
Endocardial ganglion plexus ablation (cardioneuroablation) represents a promising therapeutic technique for the treatment of vasovagal syncope (VV), functional atrioventricular block (AVB) and sinus node dysfunction (SND) with a component of vagal hypertonia. Nevertheless, there is currently a paucity of literature about the results according to the type of presentation (VV, AVB or SND). The investigators aim to assess the safety and efficacy of cardioneuroablation for the treatment of symptomatic SND.

DETAILED DESCRIPTION:
Sinus node dysfunction (SND), also known as sick sinus syndrome, comprises a wide spectrum of sinoatrial dysfunctions, ranging from sinus bradycardia, sinoatrial block, and sinus arrest to bradycardia tachycardia syndrome. An additional manifestation of SND is an inadequate chronotropic response to exercise, reported as chronotropic incompetence. Since the first cardiac denervation was reported in 2005, several registries and retrospective studies using this therapeutic approach for reflex syncope, SND and functional atrioventricular block have been published. However, due to the lack of randomized studies, current guidelines recommend permanent pacemaker implantation for patients with symptomatic SND in order to improve symptoms. Therefore, the purpose of the present study is to assess the safety and efficacy of cardioneuroablation versus permanent pacemaker implantation for the treatment of symptomatic SND.

This is a multicenter, randomized, open, interventional study. After being informed of the study and potential risks, participants will undergo a one week screening period to determine eligibility for the study entry. During this week, participants will undergo an exercise test, atropine test, and a 24 hour-holter electrocardiogram. Then, participants who meet the eligibility criteria, will be randomized 1:1 to receive permanent pacemaker implantation (control group) or cardioneuroablation (interventional group).

The primary endpoint (improve in quality of life assessed with 36-Item Short Form Survey (SF-36)) will be evaluated at six months since randomization.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic sinus node dysfunction (dizziness, asthenia or syncope) clearly related to an abnormal electrocardiogram finding (sinus arrest, sinoatrial block, extreme bradycardia (<40 bpm) or chronotropic incompetence in the exercise test).
* Absence of structural cardiopathy

Exclusion Criteria:

* Left ventricular ejection fraction <50%
* Severe valvular disease
* Any type of cardiomyopathy such as hypertrophic cardiomyopathy
* Previous ischemic heart disease
* QRS interval >130 ms
* Atrioventricular conduction disorder with a former indication of pacemaker implantation (atrioventricular block Mobitz II, advanced atrioventricular block, complete atrioventricular block)
* Lifetime expectance <12 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the SF-36 Health Survey of quality of life | Baseline and 6 months
  The SF-36 Health Survey is a validated, well known generic test for assessment of the health-related quality of life of patients.

SECONDARY OUTCOMES:
6 month free survival from permanent pacemaker implantation in the interventional group (cardioneuroablation) | Baseline and 6 months
  Percentage of patients free from pacemaker at one year in the cardioneuroablation group
Change in maximal heart rate and chronotropic incompetence in the exercise test | Baseline and 6 months
  All patients will perform a baseline exercise test and after 6 months. Maximal heart rate and chronotropic response will be recorded.
Differences in complications rates between both gropus | Baseline and 6 months
  Most common complications regarding the procedure. In the cardioneuroablation group; complications regarding vascular access and pericardial tamponade. In the pacemaker group, pneumothorax, device infection and vascular access.
Differences in 6 month free survival from syncope between both groups | Baseline and 6 months
  Syncope will be defined as any spontaneous loss of conscious with posterior recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Minguito Carazo, MD, Principal Investigator — Hospital Clinico Universitario de Santiago; Moises Rodríguez Mañero, PhD, Study Director — Hospital Clinico Universitario de Santiago; Jose Ramón González Juanatey, PhD, Study Chair — Hospital Clinico Universitario de Santiago
Locations (1):
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and informed consent form will be available for any who requires.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Baseline to 2 years

REFERENCES:
- [Background] Pachon-M JC, Pachon-M EI, Pachon CTC, Santillana-P TG, Lobo TJ, Pachon-M JC, Zerpa-A JC, Cunha-P MZ, Higuti C, Ortencio FA, Amarante RC, Silva RF, Osorio TG. Long-Term Evaluation of the Vagal Denervation by Cardioneuroablation Using Holter and Heart Rate Variability. Circ Arrhythm Electrophysiol. 2020 Dec;13(12):e008703. doi: 10.1161/CIRCEP.120.008703. Epub 2020 Nov 16. PMID 33198486
- [Background] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05186220/Prot_SAP_000.pdf